CLINICAL TRIAL: NCT06151145
Title: Stepped Care for Weight Loss Maintenance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00404188; R01NR020197 (NIH)
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Obesity
Keywords: obesity; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (Active Comparator): Usual care
  Interventions: Behavioral: Usual care
- Text-message intervention with digital tools (SELF) (Experimental): Text-message intervention
  Interventions: Behavioral: SELF
- Stepped Care (STEP) (Experimental): Stepped care
  Interventions: Behavioral: STEP

INTERVENTIONS:
Behavioral: Usual care — Participants in usual care will be emailed monthly educational modules with information on maintaining weight loss.
  Arms: Usual care
Behavioral: SELF — The SELF group will receive a wireless "smart" body weight scale and wearable physical activity tracker, and text messages.
  Arms: Text-message intervention with digital tools (SELF)
Behavioral: STEP — The STEP intervention consists of 4 steps that are progressive and based on response to treatment. Step 1: Digital health intervention. The first step will be the digital health intervention as described under SELF. Step 2: Monthly, in-person counseling. Participants who move to Step 2 will be provided with monthly, in-person counseling. Step 3: Twice per month counseling. Step 3 will be twice-monthly counseling, spaced at every other week. Step 4: Meal replacements. Participants will be prescribed a partial meal replacement program.
  Arms: Stepped Care (STEP)

SUMMARY:
This study is a 3-group, parallel design, randomized controlled trial (RCT) in approximately 258 adults with obesity that will investigate whether a 16-week behavioral weight loss treatment and a 52-week stepped-care digital health intervention can improve the maintenance of a ≥ 5% weight loss.

16-week run-in (Phase 1). To qualify for randomization, participants must lose ≥ 5% of initial weight in the 16-week run-in. This loss will be achieved with the provision of weekly-group lifestyle counseling, which includes a partial meal replacement diet.

52-week randomized trial of 3 weight loss maintenance strategies (Phase 2): Participants who have achieved ≥ 5% weight loss during Phase 1 will be randomly assigned to 1 of 3 groups:

1. Participants in the Usual Care group will be emailed monthly educational modules with information on maintaining weight loss.
2. Participants in the SELF group will receive a wireless "smart" body weight scale and a wearable physical activity tracker, and daily text messages with tailored feedback to assist in weight loss maintenance.
3. Participants in the STEP group will be enrolled in an intervention that consists of 4 steps that are progressive and based on response to treatment. After 13 weeks at each step, participants who do not maintain a ≥5% weight loss or regain 2 percentage points of weight from the participants randomization value will move to a higher intensity step. Participants who maintain weight loss will stay at the same step.

ELIGIBILITY:
Inclusion Criteria:

* BMI>/=30 kg/m2 or >/=27 kg/m2 with an obesity-related complication
* Age 18-70 years
* Completion of baseline assessment tasks
* Ability to engage in physical activity
* Own a smartphone capable of receiving text-messages and syncing to weight scales and physical activity trackers
* Home wireless access

Exclusion Criteria:

* Serious medical condition or psychiatric condition that may pose a risk to the participant during intervention, cause a change in weight, or limit ability to adhere to the behavioral recommendations of the program
* Pregnant or planning pregnancy in the next 1.5 years
* Weight>440 lbs
* Planned move out of the area in the next 1.5 years
* Recently began a course of or changed the dosage of medication that can cause significant change in weight
* History of bariatric surgery
* Weight loss of >5% in the previous 6 months
* Household member already participating in study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Weight (kg) change for STEP versus usual care | Baseline, 52 weeks
  Weight change (kg) for STEP versus usual care
Weight (kg) change for SELF versus usual care | Baseline, 52 weeks
  Weight change (kg) for SELF versus usual care

SECONDARY OUTCOMES:
Change in self-weighing frequency (days) for STEP and SELF versus usual care | Baseline, 52 weeks
  Change in number of days of self-weighing for STEP and SELF versus usual care
Change in daily calorie intake for STEP and SELF vs usual care | Baseline, 52 weeks
  Change in daily calorie intake measured using 24-hour dietary recalls for STEP and SELF versus usual care
Change in physical activity (minutes) for STEP and SELF versus usual care | Baseline, 52 weeks
  Change in self-reported minutes of physical activity for STEP and SELF versus usual care
Weight (kg) change for STEP versus SELF | Baseline, 52 weeks
  Weight change (kg) for STEP versus SELF
Change in days of self-weighing for STEP versus SELF | Baseline, 52 weeks
  Self-weighing frequency for STEP versus SELF
Change in daily calorie intake for STEP versus SELF | Baseline, 52 weeks
  Change in daily calorie intake measured using 24-hour dietary recalls for STEP versus SELF
Change in self-reported minutes of Physical activity for STEP versus SELF | Baseline, 52 weeks
  Change in self-reported minutes of physical activity for STEP versus SELF

OTHER OUTCOMES:
Cost effectiveness | Up to 52 weeks
  To evaluate the incremental cost effectiveness per unit decrease in weight (kg) from a healthcare payer perspective

CONTACTS AND LOCATIONS:
Overall Officials: Ariana M Chao, PhD, CRNP, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States